CLINICAL TRIAL: NCT07020026
Title: Evaluation of Tau-Pathology in Sporadic and LRRK2 Parkinson's Disease Using [18F]PI-2620: A High-resolution PET Imaging Study Using NeuroEXPLORER (NX PI-2160 in PD)
Brief Title: Evaluation of Tau-Pathology in Sporadic and LRRK2 Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: XI-001 (PPMI 029)
Record Dates: First submitted 2025-05-23; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — ((18)F)PI-2620

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Parkinson's Disease (PD) (Experimental): Sporadic and LRRK2
  Interventions: Drug: [18F]PI-2620
- Tauopathy (Experimental): Progressive Supranuclear Palsy (PSP) and Corticobasal Syndrome (CBS)
  Interventions: Drug: [18F]PI-2620
- Healthy (Experimental): Healthy participants
  Interventions: Drug: [18F]PI-2620

INTERVENTIONS:
Drug: [18F]PI-2620 — All participants will undergo PET imaging using the [18F]PI-2620 tau-binding tracer.

SUMMARY:
The study aims to evaluate the burden of tau pathology in people with Sporadic and LRRK2 PD via in vivo imaging using the tau tracer, [18F]PI-2620, and a high resolution PET camera, NeuroEXPLORER.

DETAILED DESCRIPTION:
The purpose of this study to compare how well [18F] PI-2620, a PET radiotracer targeting Tau protein, bind to brain regions in people with Parkinson's disease (PD), Progressive Supranuclear Palsy, Corticobasal Syndrome, and healthy volunteers.

The study is planned to be conducted over a period of two years. The study aims to assess the tau burden in PD compared to diseased and healthy controls with PET imaging using [18F]PI-2620 and utilizing the new NX PET camera. The study will include subjects already enrolled in the PPMI study to enable efficient enrollment. The study will utilize clinical and imaging assessments obtained during the PPMI study visit to reduce the subject burden and enable longitudinal PPMI study data used in the study analysis.

In the first year, half of the cohort will be recruited including 10 sporadic PD, 10 LRKK2 PD, 5 PSP/CBS, and 5 Healthy controls. The first-year cohorts, may be scanned on both the NX and the conventional PET camera to allow for comparison of tau deposits visualization between the two camera systems.

During the second year, remaining cohorts will be recruited to acquire the [18F]PI-2620 image using the NX PET camera. In order to investigate the temporal change in tau pathology in PD, participants recruited in the first year will be followed up at 12 months with repeat imaging with NX.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria include the following:

1. Ability to comply with the study procedures and attend follow-up visits.
2. Written informed consent from the participant or legal guardian.
3. Male or Female between 45 years and 85 years of age (Females must meet additional criteria specified below, as applicable) a. Females must be of non-childbearing potential or using a highly effective method of birth control 14 days prior to until at least 24 hours after injection of [18F]PI-2620 or DaTscan.

i. Non-childbearing potential is defined as a female that must be either postmenopausal (no menses for at least 12 months prior to PET scan) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).

ii. Highly effective method of birth control is defined as practicing at least one of the following: A birth control method that results in a less than 1% per year failure rate when used consistently and correctly, such as oral contraceptives for at least 3 months prior to injection, an intrauterine device (IUD) for at least 2 months prior to injection, or barrier methods, e.g., diaphragm or combination condom and spermicide. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.

b. Females of childbearing potential must not be pregnant, breastfeeding or lactating, or planning pregnancy during the duration of the study.

c. Non PPMI participant females of childbearing potential must have a negative serum pregnancy test at Screening and all females of childbearing potential must have negative urine pregnancy test prior to [18F]PI-2620 injection on day of Baseline PET scan.

d. Non PPMI participant females of childbearing potential must have a negative urine pregnancy test prior to Screening Visit DaTscan injection.

Healthy Controls:

a) Enrolled in the PPMI study as a healthy subject.

Disease specific inclusion criteria:

a) Parkinson's disease

a. Enrolled in the PPMI study as a sporadic PD or LRRK2 PD participant. b. Known CSF alpha synuclein seeding amplification assay status. c. Known Plasma phosphorylated Tau217 status. b) Progressive Supranuclear Palsy (PSP):

1. Diagnosis of progressive supranuclear palsy (PSP) based on the Clinical diagnosis of progressive supranuclear palsy: The movement disorder society criteria (Höglinger et al., 2017).
2. Symptom onset within 2-5 years prior to screening.
3. Progressive motor symptoms including vertical supranuclear gaze palsy, postural instability, and other signs of parkinsonism.
4. Evidence of striatal degeneration in form of abnormal DaTscan (previously obtained DaTscan since onset of motor symptoms may be used).

c) Corticobasal Syndrome (CBS):

1. Diagnosis of corticobasal syndrome (CBS) based on clinical criteria, with asymmetric motor and cognitive dysfunction (Armstrong et al., 2013).
2. Presence of limb apraxia, dystonia, alien limb phenomenon, and/or parkinsonism (e.g., rigidity, bradykinesia).
3. Cognitive decline as indicated by impairment in attention, executive function, or memory.
4. Evidence of striatal degeneration in form of abnormal DaTscan (previously obtained DaTscan since onset of motor symptoms may be used).

Exclusion Criteria:

1. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
2. For those receiving Screening DaTscan:

   • Received any of the following medications that could interfere with the imaging and unwilling or medically unable to hold them for five half-lives before SPECT imaging: alpha methyldopa, methylphenidate, amphetamine derivatives or modafinil, bupropion, phentermine, phencyclidine, fentanyl, or medication commonly considered to interfere with Ioflupane binding per standard clinical practice.
3. Received any of the following drugs: dopamine receptor blockers (neuroleptics), metoclopramide and reserpine, within 6 months of Screening Visit for non-PPMI participants or within 6 months of Baseline Visit for PPMI participants.
4. Any structural abnormality or finding on previously obtained or screening brain MRI suggestive of clinically significant neurological disorders other than the diseases of interest (in the opinion of the investigator).
5. Any other reason that in the opinion of the investigator, including abnormal labs, that could interfere with the safety with radiotracer injection, would render the participant unsuitable for the study enrollment.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of tau binding between study cohort using Standardized Uptake Value ratio ( SUVr) | Once during single PET imaging
  Determination of [18F]PI-2620 binding in brain regions in all participants with NX acquired images to compare tau binding between study cohorts.

SECONDARY OUTCOMES:
Comparison of Tau imaging to clinical profile | Once during single PET imaging
  To compare [18F]PI-2620 binding with clinical assessments including motor and cognitive rating scale.
Comparison of Tau imaging to biomarker profile | Once during single PET imaging
  To compare [18F]PI-2620 binding with CSF Synuclein Seed Amplification status. To compare [18F]PI-2620 binding with plasma phosphoTau217.
Compare Tau binding between Standard and high-resolution PET camera in all participants using SUVr. | Once during single PET imaging
  To compare the tau binding in all participants between the NX and conventional PET scanner (Siemens Biograph mCT).
Compare longitudinal change | 12 months
  To compare longitudinal change in [18F]PI-2620 binding over a period of 12 months across all cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Marek, MD, Study Chair — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders / XingImaging, LLC, New Haven, Connecticut, United States